CLINICAL TRIAL: NCT02686528
Title: Are Postoperative Hip Precautions Necessary After a Total Hip Arthroplasty Via the Posterior Approach: A Prospective Randomized Trial
Brief Title: Postoperative Hip Precautions After Total Hip Arthroplasty Via the Posterior Approach: A Prospective Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Omar Behery, Assistant Professor, Orthopaedic Surgery Adult Reconstruction and Replacement, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13100906
Record Dates: First submitted 2016-01-11; First posted 2016-02-19 (Estimated); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis; Degenerative Joint Disease
Keywords: total hip arthroplasty; hip precautions; posterior approach
MeSH Terms: conditions — Osteoarthritis; Joint Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Hip Precautions (Experimental): Patients will not be prescribed hip precautions in the first 6 weeks after surgery. The hip precautions that will no longer be prescribed are: no hip flexion past 90º, no crossing the legs, and no twisting at the waist.
  Interventions: Other: No Hip Precautions
- Hip Precautions (Active Comparator): Patients will receive the following hip precautions: no hip flexion past 90º, no crossing the legs, and no twisting at the waist for the first six weeks after surgery.
  Interventions: Other: Hip Precautions

INTERVENTIONS:
Other: Hip Precautions — Hip precautions are functional limitations of the hip replacement prescribed to patients for the first six weeks after surgery and are no hip flexion past 90º, no crossing the legs, and no twisting at the waist.
  Arms: Hip Precautions
Other: No Hip Precautions — Patients will not be prescribed hip precautions in the first 6 weeks after surgery. The hip precautions that will no longer be prescribed are: no hip flexion past 90º, no crossing the legs, and no twisting at the waist.
  Arms: No Hip Precautions

SUMMARY:
The purpose of this study is to determine if hip precautions, which are instructions that limit functional use of a hip replacement after surgery, affect the rate of dislocation in the first six weeks after primary total hip replacement surgery. The impact of hip precautions on a patient's return to activities of daily living and overall patient satisfaction will also be investigated. The overall cost effectiveness of hip precautions will be determined.

DETAILED DESCRIPTION:
This study examines the necessity of postoperative hip precautions in patients after primary total hip arthroplasty via the posterior approach. Precautions are instructions that limit the functional use of the hip and are given for the first six weeks after surgery, with the goal of preventing an instability event resulting in dislocation. The hip precautions that will be investigated in this study are: no hip flexion past 90º, no crossing the legs, and no twisting at the waist.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary total hip arthroplasty via the posterior approach by participating attending surgeons at this institution
* Index diagnosis of noninflammatory arthritis
* Patients must be able to understand and comply with study procedures

Exclusion Criteria:

* Allergy or intolerance to the study materials
* History of previous surgeries on the affected joint other than arthroscopy; i.e. revision THA or open surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1133 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Dislocation | 6 weeks after surgery
  Incidence of dislocation of the total hip arthroplasty will be recorded for both treatment groups.

SECONDARY OUTCOMES:
Activities of Daily Living | 1 year after surgery
  The time from surgery to return to activities of daily living will be measured for both treatment groups. This includes return to activities of bathing, return to work, and return to driving.

OTHER OUTCOMES:
Use of Assistive Devices After Surgery | 6 months after surgery
  Patients will be surveyed in clinic after surgery about their use of assistive devices including seat extenders, extra pillows between the legs, and walkers. The use of these devices between groups will be compared and the cost per patient in each group for use of these devices will be determined, allowing for analysis of potential cost savings for patients not prescribed hip precautions.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Behery, MD, Principal Investigator — Orthopedics Surgeon
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No